CLINICAL TRIAL: NCT06423365
Title: Development, Testing, and Implementation of Virtual Statin Associated Muscle Symptom Management
Brief Title: A Tool to Help Patients With Muscle Symptoms After Taking a Statin Medication.
Acronym: 1821534-10
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Kaiser Permanente (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jordan King, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1821534-10; R01HL157439 (NIH)
Record Dates: First submitted 2024-04-20; First posted 2024-05-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Hydroxymethylglutaryl-CoA Reductase Inhibitors; Hypercholesterolemia; Cardiovascular Diseases; Pharmacists; Placebo Effect
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Participants randomized to usual care will continue to receive usual care at Kaiser Permanente Colorado as they would under normal, non-study conditions.
- Usual Care + Virtual Statin Management (VSM) (Experimental): Participants randomized to usual care + virtual statin management (VSM) will continue to receive usual care at Kaiser Permanente Colorado as they would under normal, non-study conditions, and they will also be given a link to engage with the VSM website. The VSM website is an educational tool which has four principal components: 1) learning how to distinguish if and when muscle symptoms are caused by the statin; 2) learning the essentials about heart disease, focusing on causes, risk factors, and the crucial role of cholesterol management in prevention; exploring various cholesterol lowering options, including when it makes sense to retry a statin and what options exist beyond statins; and 4) learning to engage in productive discussions with healthcare providers and set effective treatment goals together.
  Interventions: Other: Virtual Statin Management (VSM)

INTERVENTIONS:
Other: Virtual Statin Management (VSM) — VSM is a web-based decision aid to help manage statin therapy after experiencing muscle pain perceived to be caused or worsened by their statin therapy. The introduction will feature a brief explanation of the tool and what they can expect. The modules are:
  1. General education (lipids, heart disease, medications)
  2. Side effects (causes, diagnosis).
  3. Statin modifications. VSM will guide patients to understand their lipid-lowering options, particularly their statin options that may best match patients' stated preferences.
  4. ASCVD risk & statin benefit. Finally, the VSM experience will end by providing the patient with a summary of the results of their use of the tool, which can be used during discussions with their healthcare provider. The information gathered from the VSM will remain confidential and will not be disclosed to anyone other than the patient.
  Arms: Usual Care + Virtual Statin Management (VSM)

SUMMARY:
The goal of this clinical trial is to learn if an educational website can help patients make an informed decision and engage in shared decision-making with their healthcare provider regarding cholesterol lowering medication use after they have stopped statin therapy due to self-reported muscle symptoms from taking a statin medication. The main questions the trial aims to answer are:

1. Compared to usual care, are patients who engage with the website after experiencing statin-associated muscle symptoms (SAMS) more likely to retry statin therapy?
2. Compared to usual care, are patients who retry statin therapy after engaging with the website more likely to persist on statin therapy?

Researchers will compare people randomized to use the website to those who are receiving usual care to see if statin re-start and persistence rates change.

All participants will take baseline questionnaires and receive usual care as they would if they were not in the study (e.g., visit their doctor, get labs drawn, take medication as prescribed). Patients randomized to the website arm will be asked to engage with content in a website which is anticipated to take most patients approximately 30-minutes. Their clinician will then contact them for a follow-up visit as needed.

ELIGIBILITY:
Inclusion Criteria:

* KPCO member
* Sold a statin from KPCO pharmacy in the previous six months
* Have a gap of >1.0x the days' supply in refilling their statin
* Patient who stopped therapy (or delayed filling prescription) due to some perceived side effect
* Has email address available in kp.org (and therefore has access to a computer with internet)

Exclusion Criteria:

* Unable to verbalize comprehension of study or impaired decision-making
* Non-English speaking
* Limited life expectancy (e.g. hospice or palliative care)
* Pregnant or planning to become pregnant
* Patients on Kaiser Permanente's "do not call" list for research will also be excluded.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 816 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who retry statin therapy | 30 days post-enrollment
  Measured using pharmacy dispensing records
Number of participants who continue to take statin therapy | 6 months post-enrollment
  Measured using pharmacy dispensing records

SECONDARY OUTCOMES:
How adherent participants are to prescribed statin therapy | 6 months post-enrollment
  Measured using pharmacy dispensing records, using the proportion of days' covered calculation metric (range: 0-100%, where 100% means perfectly adherent)

OTHER OUTCOMES:
Proportion of participants satisfied with their treatment | 6 months post-enrollment
  Assessed using two questions inspired by the Treatment Satisfaction with Medication Questionnaire. Participants the degree to which they agree or disagree (5-point Likert) regarding their satisfaction with cholesterol-lowering medication.
Participant-reported decisional conflict | 1 month post-enrollment
  Assessed using the Decisional Conflict Scale, 10-item, 3-response (https://decisionaid.ohri.ca/docs/develop/Tools/DCS_LowLiteracy_English.pdf). Participants indicate "yes", "unsure", or "no" to 10 questions assessing their decisional conflict regarding their decision to use cholesterol-lowering medication.
Participant-reported decision self-efficacy | 6 months post-enrollment
  Measured using the Decision Self-Efficacy Scale, 11-item, 3-response (https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decision_SelfEfficacy.pdf). Participants indicate their level of confidence from 0 (not at all confident) to 4 (very confident) regarding their decision to use cholesterol-lowering medication.
Participant-reported perception of cardiovascular disease risk | 6 months post-enrollment
  Adapted from 3 questions used in the Prospective Assessment of Lipid Management (PALM) registry (https://classic.clinicaltrials.gov/ct2/show/NCT02341664). Participants indicate their perceived risk for having a heart disease event.
Participant-reported degree of trust in healthcare | 6 months post-enrollment
  Measured using the Trust in Physician Scale, 11-item (https://pubmed.ncbi.nlm.nih.gov/2084735/). Participants indicate the degree to which they agree or disagree (5-point Likert scale) with statements regarding their trust in healthcare personnel.
Participant-reported statin conspiracy beliefs | 6 months post-enrollment
  Participants indicate the degree to which they agree or disagree with 18 statements regarding potential statin-related harms or conspiracies. Answer options of strongly disagree, disagree, neither agree nor disagree, agree, strongly agree, or Not sure. Agreement with the statement indicates a negative belief about statins.
Participant-reported decision regret | 6 months post-enrollment
  Measured using the Decision Regret Scale, 5-item, 5-response (https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Regret_Scale.pdf). Participant indicate the degree to which they agree or disagree (5-point Likert Scale) with 5 statements regarding their choice to use cholesterol-lowering medication.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan B King, PharmD, MS, Principal Investigator — University of Utah
Locations (1):
- Kaiser Permanente Colorado, Aurora, Colorado, United States